CLINICAL TRIAL: NCT01236586
Title: A Phase 1/2 Study of RO4929097, An Oral Small Molecule Inhibitor of Gamma-Secretase, in Children With Relapsed/Refractory Solid or CNS Tumors, Lymphoma, or T-Cell Leukemia
Brief Title: RO4929097 in Children With Relapsed/Refractory Solid or CNS Tumors, Lymphoma, or T-Cell Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: CTEP/National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110017; 11-C-0017
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-13

CONDITIONS: Lymphoma; Brain Neoplasms; Sarcoma; Osteosarcoma; Wilm's Tumor
Keywords: Maximum Tolerated Dose; Toxicity; Pharmacokinetics; NOTCH Signaling Pathway; Expression of JAGGED 1 and 2; Cancer; Solid Tumor; Brain Tumor; Wilms Tumor; Osteosarcoma; Lymphoma
MeSH Terms: conditions — Lymphoma; Brain Neoplasms; Sarcoma; Osteosarcoma; Wilms Tumor; Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Dexamethasone

INTERVENTIONS:
Drug: RO4929097
Drug: Dexamethasone

SUMMARY:
Background:

- The anti-cancer drug RO4929097 is being tested for its ability to block blood vessel growth to tumors and slow or stop the growth of cancer cells. However, it has been used in only a small number of adults and has not yet been tested in children. Researchers are interested in determining whether RO4929097 is a safe and effective treatment for tumors or leukemia that has not responded to standard treatment.

Objectives:

- To determine the safety and effectiveness of RO4929097 as a treatment for children and adolescents who have been diagnosed with certain kinds of cancer that have not responded to standard treatment.

Eligibility:

- Children, adolescents, and young adults between 1 and 21 years of age who have been diagnosed with solid, nervous system, or blood-based cancers that have not responded to standard treatment.

Design:

* Participants will be screened with a medical history, physical examination, blood and urine tests, and imaging studies. Some participants may also have a bone marrow biopsy to evaluate the state of their disease.
* Participants will be separated into three groups: One group will receive RO4929097 alone, and the other two will receive RO4929097 in combination with the immune-suppressing drug dexamethasone.
* RO4929097 will be given as tablets on one of two schedules: days 1 to 3 of every week (Schedule A) or days 1 to 5 of every week (Schedule B). The dosing schedule will be determined randomly. Every 4-week treatment period is one cycle, and participants may receive RO4929097 for up to 24 cycles.
* Participants will have frequent blood and urine tests and imaging studies to evaluate the progress of treatment, and will be asked to keep a diary to monitor any side effects.

DETAILED DESCRIPTION:
Background:

* Notch signaling is aberrantly activated in a variety of human tumors including solid tumors and hematological malignancies including T-cell leukemia (T-ALL) and pediatric cancers, such as osteosarcoma, gliomas, medulloblastomas, ependymoma, and hematological malignancies.
* One emerging strategy to inhibit Notch signaling is the use of gamma-secretase inhibitors (GSIs), which prevent Notch receptor activation cleavage.
* RO4929097 is an orally administered small molecule that is a potent and selective GSI, which has shown antitumor activity in preclinical studies.

Objectives:

* To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose, and associated toxicities of RO4929097 administered orally to children with relapsed/refractory solid tumors or lymphoma on 2 schedules: once daily orally on a 3 day on/4 day off weekly schedule (schedule A) and once daily for 5 consecutive days weekly schedule (schedule B).
* To determine the MTD and recommended Phase 2 dose, and associated toxicities of RO4929097 administered with dexamethasone.
* To characterize the pharmacokinetics of RO4929097 in children with refractory cancer.
* To preliminarily define the anti-tumor activity of RO4929097 in children with refractory solid tumors within the confines of a phase I study.
* To determine initial efficacy on the anti-tumor activity of RO4929097 when combined with dexamethasone in children with relapsed/refractory T-ALL.
* To study the effects of RO4929097 on components of the Notch signaling pathway in peripheral blood mononuclear cells and/or T-ALL blasts, to examine archival tumor samples for expression or amplification of target molecules, and to preliminarily assess changes after treatment using FDG PET imaging.

Eligibility:

* Patients greater than 12 months and less than or equal to 21 years of age with a diagnosis and histologic verification (except patients with intrinsic brain stem tumors, optic pathway gliomas) of measureable or evaluable relapsed or refractory disease. Current disease state must be one for which there is no known curative therapy, or therapy proven to prolong survival with an acceptable quality of life.
* Subjects must be able to swallow tablets.
* Patients who are pregnant, are known to be serologically positive for Hepatitis A, B, C, or have a history of liver disease, or have prolonged QTc are not eligible.

Design:

* This phase I study will first evaluate the safety and pharmacokinetics of RO4929097 administered orally to children with relapsed/refractory solid tumors (Part 1) on 2 schedules: once daily on a 3 day on/4 day off weekly schedule (Schedule A) and once daily for 5 consecutive days weekly schedule (Schedule B).
* One cycle will be 28 days, and subjects may continue cycles in the absence of progressive disease or unacceptable treatment-related toxicity to a total of 24 cycles.
* After determining MTD of RO4929097, an evaluation of RO4929097 plus concomitant dexamethasone (Part 2) in at least one of the schedules tested in Part 1, will be undertaken.
* After the MTD of RO4929097 plus dexamethasone has been identified, enrollment of subjects with relapsed/refractory T-ALL (Part 3) will be undertaken to obtain initial efficacy data in this patient population.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Patients greater than 12 months and less than or equal to 21 years of age with a diagnosis and histologic verification (except patients with intrinsic brain stem tumors, optic pathway gliomas) of measureable or evaluable relapsed or refractory disease. Current disease state must be one for which there is no known curative therapy, or therapy proven to prolong survival with an acceptable quality of life.
* Subjects must be able to swallow tablets.
* Patients who are pregnant, are known to be serologically positive for Hepatitis A, B, C, or have a history of liver disease, or have prolonged QTc are not eligible.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10-08; Primary Completion 2011-04-13 (Actual); Study Completion 2011-04-13 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of this study are self-reported fatigue, depression, and quality of life scores of patients before, at midpoint, and at completion of each cycle of their cancer treatment.

SECONDARY OUTCOMES:
Cytokine profile

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - St. Jude Childrens Research Hospital, Memphis, Tennessee

REFERENCES:
- [Background] Artavanis-Tsakonas S, Rand MD, Lake RJ. Notch signaling: cell fate control and signal integration in development. Science. 1999 Apr 30;284(5415):770-6. doi: 10.1126/science.284.5415.770. PMID 10221902
- [Background] Curry CL, Reed LL, Golde TE, Miele L, Nickoloff BJ, Foreman KE. Gamma secretase inhibitor blocks Notch activation and induces apoptosis in Kaposi's sarcoma tumor cells. Oncogene. 2005 Sep 22;24(42):6333-44. doi: 10.1038/sj.onc.1208783. PMID 15940249
- [Background] Bray SJ. Notch signalling: a simple pathway becomes complex. Nat Rev Mol Cell Biol. 2006 Sep;7(9):678-89. doi: 10.1038/nrm2009. PMID 16921404